CLINICAL TRIAL: NCT03231150
Title: Randomized Clinical Study to Evaluate Ultrasound Guided Injection Therapy Versus Topographic Injection Therapy for Plantar Fasciitis
Brief Title: Plantar Fasciitis Randomized Clinical Control Trial
Acronym: PF-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PPMC-04
Record Dates: First submitted 2017-07-21; First posted 2017-07-27 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Plantar Fascitis

STUDY DESIGN:
Intervention Model Description: This investigation will be chronologically divided into four stages that will commence after procurement of institutional review board (IRB) approval and funding, namely: 1) screening and enrollment, 2) random treatment allocation and treatment, 3) data collection and analysis, and 4) presentation and publication. We anticipate that it will take approximately 23.5 months to execute the clinical experiment and to prepare the report for publication.
Who Masked: Care Provider, Investigator
Masking Description: Participants that do not experience at least a 50% reduction in pain following phase 1 will undergo randomization to either USGI or ATGI, both injections consisting of 0.5 ml 0.25% bupivacaine plain, 0.5 ml dexamethasone phosphate, and 0.5 ml triamcinolone acetonide 40 mg/ml. Execution of the USGI will employ an actual diagnostic US machine (Voluson E8 Expert, General Electric Company, Boston, MA) and a plantarmedial approach, whereas execution of the ATGI will employ a sham diagnostic US machine and a plantarmedial approach. The patients will be randomized into these groups by a specialized statistical computerized system that randomly selects a number to the participant. An even or an odd number represents which form of injection the patient is to receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anatomical injection (Active Comparator): Once patient has been randomized, if placed in the anatomically-guided injection group, the medial band of the plantar fascia origin on the calcaneus will be palpated and marked approximately. In the clinical setting, a sham ultrasound machine will be utilized to "locate" the plantar fascia keeping the patient blinded to the treatment modality. The area will then be prepped with alcohol to the medial heel and utilizing a medial approach, an injection of 0.5 cc 0.5% bupivacaine, 0.5 cc dexamethasone and 0.25 cc triamcinolone acetamide 40 mg/mL will be administered into the area surrounding the plantar fascia. The area will then be cleaned will alcohol and dressed with a small elastic bandage.
  Interventions: Procedure: Local Steroid Injection into the plantar heel; Procedure: Anatomical Guided injection
- Ultrasound Guided Injection (Experimental): Once patient has been randomized, if placed in the USGI group, the patient will be scheduled for an ultrasound therapy in the radiology department at Penn Presbyterian Medical Center. In this setting, the patient will be informed that in order to keep them blinded, that all patients must have either injection performed in the radiology department and that the ultrasound machine utilized will either be on or off during the injection keeping the patient blinded to the treatment modality. The area will then be prepped with alcohol to the medial heel and utilizing a medial approach, an injection of 0.5 cc 0.5% bupivacaine, 0.5 cc dexamethasone and 0.25 cc triamcinolone acetamide 40 mg/mL will be administered into the area surrounding the plantar fascia. The area will then be cleaned will alcohol and dressed with a small elastic bandage.
  Interventions: Procedure: Local Steroid Injection into the plantar heel; Procedure: Ultrasound Guided Injection

INTERVENTIONS:
Procedure: Local Steroid Injection into the plantar heel — Injections consisting of 0.5 ml 0.25% bupivacaine plain, 0.5 ml dexamethasone phosphate, and 0.5 ml triamcinolone acetonide 40 mg/ml.
Procedure: Ultrasound Guided Injection — Execution of the USGI will employ an actual diagnostic US machine (Voluson E8 Expert, General Electric Company, Boston, MA) and a plantarmedial approach
  Arms: Ultrasound Guided Injection
Procedure: Anatomical Guided injection — Execution of the ATGI will employ a sham diagnostic US machine and a plantarmedial approach.
  Arms: Anatomical injection

SUMMARY:
The primary aim of this clinical experiment is to compare, in terms of pain relief measured using the 10-cm visual analog scale (VAS) pain score (5-7), the clinical results of ultrasound-guided injection (USGI) versus anatomic topography-guided injection (ATGI) of corticosteroid for the treatment of proximal PF. Secondary aims will be to compare foot-related quality of life, as measured using the Foot Function Index (FFI)and the Bristol Foot Score (BFS), between the injection groups, and also to compare the pre-injection to late-term post-injection thickness of the plantar fascia as measured in the nested USGI group.

DETAILED DESCRIPTION:
Clinically, proximal PF causes plantar heel pain, which may extend into the proximal portion of the plantar longitudinal arch. Typically, the pain is most notable upon initial weight bearing ambulation (post-static dyskinesia, PSD), such as the first step in the morning or following a period of non-weight bearing or rest. This can be attributed to walking on hard surfaces or barefoot, prolonged weight bearing activity, inadequate stretching and use of poor footwear, as well as increased amounts of walking. Standard treatment of PF includes the use of foot orthotics, both pre-fabricated and custom molded, physical therapy and myotendinous stretching, splinting or strapping the foot, nonsteroidal anti-inflammatory drugs, ice, and corticosteroid injections. Ultrasonography (US) can be useful for examining the plantar fascia, which typically measures between 2 mm to 4 mm in thickness, and findings indicative of PF include diffuse hypoechogenicity at the calcaneal attachment of the plantar fascia, loss of definition between the plantar fascia and the surrounding soft tissues, peri-insertion edema, and thickness over 4.5 mm. Local infiltration of corticosteroids has been used to treat PF since the 1950s. Despite this being a well established treatment, there are still unexamined features of this form of intervention, including the method of injection, type of steroid used, concurrent use of localanesthetic agents, concurrent use of orthoses and/or supportive arch strapping, concurrent physical therapy, and the use of ultrasonographic guidance of the corticosteroid injection. The primary aim of this clinical experiment is to compare, in terms of pain relief measured using the 10-cm visual analog scale (VAS) pain score (5-7), the clinical results of ultrasound-guided injection (USGI) versus anatomic topography-guided injection (ATGI) of corticosteroid for the treatment of proximal PF. Secondary aims will be to compare foot-related quality of life, as measured using the Foot Function Index (FFI)and the Bristol Foot Score (BFS), between the injection groups, and also to compare the pre-injection to late-term post-injection thickness of the plantar fascia as measured in the nested USGI group.

ELIGIBILITY:
Inclusion Criteria:

* Pain on palpation along the proximal plantar fascia with or without radiographic evidence of a plantar calcaneal bone spur
* ≥18 years of age
* Male or non-pregnant female of any ethnicity or race
* Active, former or non smoker
* With or without peripheral vascular disease without lower extremity intermittent claudication or rest pain
* With or without diabetes mellitus without polyneuropathy
* With or without collagen vascular disease without lower extremity wound formation.

Exclusion Criteria:

* Known drug or alcohol dependence
* Chronic pain syndrome or lumbosacral radiculitis
* Neurological condition that requires the use of analgesic medications or anti-seizure or neuroleptic medications
* Peripheral vascular disease that results in rest pain or intermittent claudication or venous stasis ulceration
* Calcaneal stress fracture or show evidence of a foreign body or tumor of the affected heel as viewed radiographically
* Pregnant females
* Known allergy to any of the components of the injection therapy
* Previously suffered a rupture or surgery of the plantar fascia within the 5 years preceding participation in the investigation
* Existing or prior osteomyelitis of the involved calcaneus
* Unable to consent to participation in clinical research or currently be involved in another clinical investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2017-03-28 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in VAS pain score at post injection periods with use of USGI | Baseline to 3 months, 6 month, 9 month, and 12 month follow up
  with the primary efficacy endpoint being the 3-month post injection pain score
Change in VAS pain score at post injection periods with use of ATGI | Baseline to 3 months, 6 month, 9 month, and 12 month follow up
  with the primary efficacy endpoint being the 3-month post injection pain score

SECONDARY OUTCOMES:
Observation of normal plantar fascia after treatment as measured by ultrasound (US) | Baseline to 12 month follow up
Foot-related quality of life outcomes as measured with use of the FFI | Baseline to 3 months, 6 month, 9 month, and 12 month follow up
Foot-related quality of life outcomes as measured with use of the BFS | Baseline to 3 months, 6 month, 9 month, and 12 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Donald S Malay, DPM, Principal Investigator — Penn Presbyterian Medical Center
Locations (1):
- Penn Presbyterian Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ang TW. The effectiveness of corticosteroid injection in the treatment of plantar fasciitis. Singapore Med J. 2015 Aug;56(8):423-32. doi: 10.11622/smedj.2015118. PMID 26311907
- [Result] Weil L Jr, Glover JP, Weil LS Sr. A new minimally invasive technique for treating plantar fasciosis using bipolar radiofrequency: a prospective analysis. Foot Ankle Spec. 2008 Feb;1(1):13-8. doi: 10.1177/1938640007312318.. PMID 19825686
- [Result] Young CC, Rutherford DS, Niedfeldt MW. Treatment of plantar fasciitis. Am Fam Physician. 2001 Feb 1;63(3):467-74, 477-8. PMID 11272297
- [Result] Buchbinder R. Clinical practice. Plantar fasciitis. N Engl J Med. 2004 May 20;350(21):2159-66. doi: 10.1056/NEJMcp032745. No abstract available. PMID 15152061
- [Result] Wessel J. The reliability and validity of pain threshold measurements in osteoarthritis of the knee. Scand J Rheumatol. 1995;24(4):238-42. doi: 10.3109/03009749509100881. PMID 7481589
- [Result] Lundeberg T, Lund I, Dahlin L, Borg E, Gustafsson C, Sandin L, Rosen A, Kowalski J, Eriksson SV. Reliability and responsiveness of three different pain assessments. J Rehabil Med. 2001 Nov;33(6):279-83. doi: 10.1080/165019701753236473. PMID 11766958
- [Result] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Result] Budiman-Mak E, Conrad KJ, Roach KE. The Foot Function Index: a measure of foot pain and disability. J Clin Epidemiol. 1991;44(6):561-70. doi: 10.1016/0895-4356(91)90220-4. PMID 2037861
- [Result] Barnett S, Campbell R, Harvey I. The Bristol Foot Score: developing a patient-based foot-health measure. J Am Podiatr Med Assoc. 2005 May-Jun;95(3):264-72. doi: 10.7547/0950264. PMID 15901814
- [Result] Tsai WC, Wang CL, Tang FT, Hsu TC, Hsu KH, Wong MK. Treatment of proximal plantar fasciitis with ultrasound-guided steroid injection. Arch Phys Med Rehabil. 2000 Oct;81(10):1416-21. doi: 10.1053/apmr.2000.9175. PMID 11030509
- [Result] Tsai WC, Hsu CC, Chen CP, Chen MJ, Yu TY, Chen YJ. Plantar fasciitis treated with local steroid injection: comparison between sonographic and palpation guidance. J Clin Ultrasound. 2006 Jan;34(1):12-6. doi: 10.1002/jcu.20177. PMID 16353228
- [Result] Chen CM, Chen JS, Tsai WC, Hsu HC, Chen KH, Lin CH. Effectiveness of device-assisted ultrasound-guided steroid injection for treating plantar fasciitis. Am J Phys Med Rehabil. 2013 Jul;92(7):597-605. doi: 10.1097/PHM.0b013e318278a831. PMID 23221670
- [Result] Li Z, Xia C, Yu A, Qi B. Ultrasound- versus palpation-guided injection of corticosteroid for plantar fasciitis: a meta-analysis. PLoS One. 2014 Mar 21;9(3):e92671. doi: 10.1371/journal.pone.0092671. eCollection 2014. PMID 24658102